CLINICAL TRIAL: NCT07371871
Title: A Prospective, Single-arm, Exploratory Study of Trifluridine/Tipiracil (TAS-102) Combined With Apatinib as Third-line Therapy for Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Xiaojing, Chief Physician., Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LLYJ-0022
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Advanced Gastric Cancer; TAS-102; Apatinib
MeSH Terms: interventions — Trifluridine; tipiracil; trifluridine tipiracil drug combination; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research group (Experimental)
  Interventions: Drug: Trifluridine/Tipiracil (TAS-102) combined with Apatinib

INTERVENTIONS:
Drug: Trifluridine/Tipiracil (TAS-102) combined with Apatinib — TAS-102: 35 mg/m2/dose, taken orally within 1 hour after breakfast and dinner, twice daily, on days 1-5 of each cycle, followed by a 9-day drug-free interval, with 28 days constituting one cycle.
  Apatinib: 500 mg/dose, once daily, administered continuously for 5 days followed by a 2-day break, with 28 days as one cycle. Imaging evaluation should be performed every 2-3 cycles until disease progression or intolerance occurs.

SUMMARY:
To evaluate the efficacy and safety of trifluridine/tipiracil (TAS-102) combined with apatinib as third-line therapy for advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer confirmed by histopathological or cytological diagnosis;
* unresectable locally advanced or recurrent/metastatic gastric cancer;
* age 18-75 years, regardless of gender;
* ECOG score 0-2;
* previously received second-line treatment for advanced gastric cancer with disease progression during or after treatment;
* at least one measurable lesion present according to RECIST 1.1 criteria;
* laboratory tests meeting the following requirements: (1) Blood routine: HGB≥70g/L; WBC≥4.0×10^9/L; NEUT≥1.5×10^9/L; PLT≥90×10^9/L; (2) Blood biochemistry: ALT, AST≤2.5×upper limit of normal (ULN), serum creatinine≤1.5×upper limit of normal;
* negative pregnancy test for patients of childbearing potential and voluntary use of effective and reliable contraception during the trial.

Exclusion Criteria:

* Participation in other anti-tumor drug clinical trials within 4 weeks prior to enrollment;
* Any of the following conditions that may interfere with oral medication: inability to swallow, chronic diarrhea, or intestinal obstruction;
* Concurrent receipt of any other systemic anti-tumor therapy (excluding local treatment);
* Previous treatment with VEGFR inhibitors (excluding ramucirumab; pan-targeted TKIs are excluded);
* Known history of allergy to any component of the study drugs;
* Subjects with active infectious diseases;
* Patients deemed unsuitable for enrollment by the investigator due to potential increased study-related risks or possible interference with interpretation of study results, as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate，ORR | Perform imaging evaluation At the end of Cycle 2 or Cycle3 (each cycle is 28 days).

SECONDARY OUTCOMES:
Duration of Response，DOR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
Progression-Free Survival，PFS | From date of first dose administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.

IPD SHARING:
Plan to Share IPD: Undecided